CLINICAL TRIAL: NCT01400230
Title: Diagnostic Performances of the Computed Tomographic Coronary Angiography and IntraVascular UltraSound to Evaluate Ischemia Causing Coronary Artery Stenosis
Brief Title: Diagnostic Performances of Computed TomographIc Coronary Angiography and Intravascular Ultrasound
Acronym: IMAGES-FFR
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Inje University (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Associate professor, Seoul National University Hospital
Other Study IDs: IB-2-1010-049
Record Dates: First submitted 2011-07-15; First posted 2011-07-22 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Diagnosis Coronary Artery Disease
Keywords: computed tomography; intravascular ultrasound; coronary stenosis; fractional flow reserve
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CCTA-IVUS-FFR: Patients suspected ischemic heart disease by the symptom and CCTA and undergone IVUS and FFR in the Cath Lab with CAG enrolled consecutively.
  Interventions: Procedure: diagnostic procedures CCTA, CAG, IVUS and FFR

INTERVENTIONS:
Procedure: diagnostic procedures CCTA, CAG, IVUS and FFR — Diagnostic procedures including computed tomography, coronary angiography, intravascular ultrasound, fractional flow reserve were performed in the patients suspected ischemic heart disease.
  Other Names: CCTA, Aquillion, Toshiba; IVUS, InVision Gold, Volcano and I-Lab, Boston; FFR, Pressure Wire, St.Jude medical

SUMMARY:
Diagnostic purposes of the coronary angiography is to detect stenosis (anatomy) and to detect ischemia related stenosis (function). Coronary angiography (CAG) is a gold standard invasive techniques, but has several limitations. Intravascular ultrasound (IVUS) provides tomographic intra-luminal images. Coronary computed tomographic angiography (CCTA) is helpful to assess precise anatomical information. Optimal functional criteria and their accuracy of IVUS and CCTA by fraction flow reserve (FFR) have not been compared yet.

DETAILED DESCRIPTION:
Correlation between CCTA, IVUS and FFR will be evaluated. The presence of myocardial ischemia will be assessed by fractional flow reserve (FFR).

Diagnostic performance (sensitivity, specificity, positive predictive/negative predictive values and diagnostic accuracy) of each modality will be assessed and compared.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting chest pain suspected stable angina or unstable angina
* patients permit informed consents
* patients performed all the procedures including CCTA, IVUS and FFR and present coronary artery stenosis

Exclusion Criteria:

* acute myocardial infarction
* ejection fraction less than 40%
* infarct related artery
* chronic renal insufficiency
* left main stenosis, in-stent restenosis and grafted vessels
* allergy in contrast agent and adenosine
* unable to get a informed consents

Ages: 20 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who underwent CCTA, IVUS and FFR Stable clinical condition
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2008-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 1 day
  Evaluate and compare the diagnostic accuracy of the CCTA, IVUS and angiographic parameters for the prediction of myocardial ischemia (FFR<0.8)
  1. CCTA: % area stenosis
  2. IVUS: minimum lumen area
  3. Angiography: % diameter stenosis
  Diagnostic accuracy of each parameter: (true positive+true negative)/total cases

CONTACTS AND LOCATIONS:
Overall Officials: Joon Hyung Doh, MD, PhD, Study Director — Inje University Ilsan Paik Hospital; Bon-Kwon Koo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Nam CW, Yoon HJ, Cho YK, Park HS, Kim H, Hur SH, Kim YN, Chung IS, Koo BK, Tahk SJ, Fearon WF, Kim KB. Outcomes of percutaneous coronary intervention in intermediate coronary artery disease: fractional flow reserve-guided versus intravascular ultrasound-guided. JACC Cardiovasc Interv. 2010 Aug;3(8):812-7. doi: 10.1016/j.jcin.2010.04.016. PMID 20723852
- [Result] Nam CW, Hur SH, Cho YK, Park HS, Yoon HJ, Kim H, Chung IS, Kim YN, Kim KB, Doh JH, Koo BK, Tahk SJ, Fearon WF. Relation of fractional flow reserve after drug-eluting stent implantation to one-year outcomes. Am J Cardiol. 2011 Jun 15;107(12):1763-7. doi: 10.1016/j.amjcard.2011.02.329. Epub 2011 Apr 8. PMID 21481828
- [Result] Ahn JM, Kang SJ, Mintz GS, Oh JH, Kim WJ, Lee JY, Park DW, Lee SW, Kim YH, Lee CW, Park SW, Moon DH, Park SJ. Validation of minimal luminal area measured by intravascular ultrasound for assessment of functionally significant coronary stenosis comparison with myocardial perfusion imaging. JACC Cardiovasc Interv. 2011 Jun;4(6):665-71. doi: 10.1016/j.jcin.2011.02.013. PMID 21700253
- [Result] Ben-Dor I, Torguson R, Gaglia MA Jr, Gonzalez MA, Maluenda G, Bui AB, Xue Z, Satler LF, Suddath WO, Lindsay J, Pichard AD, Waksman R. Correlation between fractional flow reserve and intravascular ultrasound lumen area in intermediate coronary artery stenosis. EuroIntervention. 2011 Jun;7(2):225-33. doi: 10.4244/EIJV7I2A37. PMID 21646065